CLINICAL TRIAL: NCT02300610
Title: A Phase I/1b Study of Enzalutamide in Combination With Gemcitabine and Cisplatin in Bladder Cancer
Brief Title: Enzalutamide in Combination With Gemcitabine and Cisplatin in Bladder Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17924
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-06

CONDITIONS: Bladder Cancer; Carcinoma, Transitional Cell; Renal Pelvis Cancer; Ureter Cancer; Urethra Cancer
Keywords: Ureteral Diseases; Urinary Bladder Diseases; Transitional Cell Carcinoma; Bladder; Carcinoma; Renal; Pelvis; Ureter; Urethra
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Ureteral Neoplasms; Urethral Neoplasms; Ureteral Diseases; Urinary Bladder Diseases; Carcinoma | interventions — enzalutamide; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Experimental): Dose Escalation: Begin with Level 1 dose of enzalutamide (orally), with standard doses of cisplatin and gemcitabine via intravenous (IV).
  Interventions: Drug: Enzalutamide; Drug: Cisplatin; Drug: Gemcitabine
- Dose Expansion (Experimental): Dose Expansion: Enzalutamide at recommended dose level with standard doses of cisplatin and gemcitabine.
  Interventions: Drug: Enzalutamide; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Enzalutamide — Enzalutamide orally once a day. Dose Escalation Level 1: 80 mg; Level 2: 160 mg. Dose Expansion at recommended dose level, after dose escalation.
  Other Names: MDV3100; XTANDI®
Drug: Cisplatin — Cisplatin at 70 mg/m^2 IV on day 1, repeated every 21 days for total of 6 cycles.
  Other Names: Platinol®; Platinol®-AQ
Drug: Gemcitabine — Gemcitabine at 1000 mg/m^2 IV on days 1, 8, repeated every 21 days for total of 6 cycles.
  Other Names: Gemzar ®

SUMMARY:
The main purpose of this study is to find out the dose of enzalutamide that can be safely given with gemcitabine and cisplatin in patients with advanced bladder cancer. Researchers also want to find out the side effects of these drugs when given together. This study will also help in finding out the effect on tumor of the combination of enzalutamide, gemcitabine and cisplatin.

DETAILED DESCRIPTION:
For the phase 1 dose escalation phase, the starting dose of enzalutamide will be 80 mg orally once a day (Level 1). The dosing regimen of cisplatin and gemcitabine will be at standard doses of Gemcitabine at 1000 mg/m^2 IV on days 1, 8 and cisplatin at 70 mg/m2 IV on day 1, repeated every 21 days for total of 6 cycles.

Three patients will be treated dose level 1 (enzalutamide 80 mg daily). If 0 patients experience dose limiting toxicity (DLT), dose escalation will be done to level 2 of enzalutamide 160 mg daily. If 1 patient experiences DLT, 3 more patients will be treated at the same dose level; if 1 of 6 experiences DLT, escalate the dose to next level, and if 2 or more of 6 experiences DLT, the dose level 1 (80 mg enzalutamide) will be the recommended dose for dose expansion cohort.

The cohort expansion will then be done by enrolling 12 patients with stage IV bladder cancer, who express androgen receptor (AR) staining of 1+ and above by immunohistochemistry (IHC), to determine the safety and tolerability of cisplatin and gemcitabine with the recommended dose level of enzalutamide (80 mg or 160 mg, depending upon the safety results from dose escalation part) in this expanded cohort of patients with AR + bladder cancer.

Enzalutamide would be continued after completion of 6 cycles of gemcitabine-cisplatin for patients exhibiting a response or stable disease, until they experience disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed evidence of transitional cell carcinoma of bladder, renal pelvis, ureter or urethra.
* Patients with Stage IV (locally advanced or metastatic) disease. Must have measurable disease, as per Response Evaluation Criteria in Solid Tumors (RECIST).
* Minimum of 4 weeks since any major surgery, completion of radiation.
* Prior treatment with cytotoxic chemotherapy is not a requirement, but allowed only if used in neoadjuvant, adjuvant or for bladder preserving protocols, as long as was administered > 6 months prior to starting study.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Life expectancy 12 weeks or more.
* Must have normal organ and marrow function.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days of the administration of the first study treatment. Women must not be lactating.
* Sexually active women of childbearing age and men should be willing to follow birth control guidelines.
* Should be able to swallow enzalutamide and comply with study requirements.

Exclusion Criteria:

* Prior treatment with any cytotoxic chemotherapy in metastatic setting. Prior treatment with cytotoxic chemotherapy is allowed only if used in neoadjuvant, adjuvant or for bladder preserving protocols, as long as was administered > 6 months prior to starting study.
* Have undergone major surgery within 4 weeks prior to study enrollment.
* Chronic treatment with steroids or any other immunosuppressant drugs.
* Should not receive immunization with attenuated live vaccines during study period or within 1 week of study entry.
* History of seizures, predisposing factors for seizures, including underlying brain injury with loss of consciousness within previous 12 months, transient ischemic attack within previous 12 months, cerebral vascular accident or brain arteriovenous malformation.
* Untreated brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
* Congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block or a history of acute myocardial infarction within the 6 months preceding enrollment.
* Known history of HIV.
* Have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study.
* Women who are pregnant or breast feeding, or women/men able to conceive and unwilling to practice birth control guidelines.
* Concurrent medications which strongly inhibit or induce CYP enzymes (gemfibrozil, Rifampin, carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, rifapentine, bosentan, efavirenz, etravirine, modafinil, nafcillin, St. John's Wort).
* History of stage III or greater cancer, except basal or squamous cell skin cancers adequately treated or any other stage I or II cancer adequately treated and disease-free for ≥ 2 years. Incidental findings of stage I or II prostate cancer that is considered to be cured with radical cystoprostatectomy is allowed.
* Prior use of enzalutamide.
* Radiation therapy via external beam or brachytherapy within 28 days of registration.
* Patients who are ineligible to receive cisplatin: Creatinine clearance of less than 60 mL/minute, hearing loss of 25 decibel (dB) at 2 contiguous frequencies, grade 2 or higher peripheral neuropathy, or New York Heart Association Class III or higher heart failure.
* Allergy/sensitivity to any study drug (gemcitabine, cisplatin, enzalutamide), or drugs chemically related to study drug, or excipients.
* Brain metastases (including treated or stable brain metastases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2019-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jingsong Zhang, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Shilpa Gupta, M.D., Study Chair — University of Minnesota Masonic Cancer Center
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Minnesota, Masonic Cancer Center, Minneapolis, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Moffitt Cancer Center and the University of Minnesota Masonic Cancer Center, February 2015 through August 2017.
Groups:
- Dose Escalation: Level 1 Dose: Dose Escalation: Level 1 dose of 80 mg enzalutamide (orally), with standard doses of cisplatin and gemcitabine via intravenous (IV).
- Dose Escalation- Level 2 Dose: Dose Escalation: Level 2 dose of 160 mg enzalutamide (orally), with standard doses of cisplatin and gemcitabine via intravenous (IV).
- Dose Expansion: Enzalutamide at MTD (160 mg) with standard doses of cisplatin and gemcitabine.
Period: Overall Study
Arm/Group | Dose Escalation: Level 1 Dose | Dose Escalation- Level 2 Dose | Dose Expansion
Started | 3 | 3 | 4
Completed | 2 | 3 | 3
Not Completed | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- Dose Escalation: Level 2 Dose: Dose Escalation: Level 2 dose of 160 mg enzalutamide (orally), with standard doses of cisplatin and gemcitabine via intravenous (IV).
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: Level 1 Dose | Dose Escalation: Level 2 Dose | Dose Expansion | Total
Number analyzed (Participants) | 3 | 3 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 2 | 5
  >=65 years | 1 | 2 | 2 | 5
Age, Continuous [Mean (Full Range); unit: years] | 65 [58 to 75] | 66.6 [56 to 75] | 65 [60 to 73] | 65.5 [56 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1
  Male | 3 | 3 | 3 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 3 | 3 | 4 | 10
  Black or African American | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Hispanic or Latino | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Recommended Dose of Enzalutamide
Description: Dose Escalation. Maximum Tolerated Dose (MTD) of Enzalutamide when given with Cisplatin and Gemcitabine at standard doses. Dose Level 1: 80 mg Enzalutamide; Dose Level 2: 160 mg Enzalutamide.
  Dose-Limiting Toxicity (DLT) is defined as any of the following occurring in the first 21 days (cycle 1) of study participation that are considered at least possibly related to enzalutamide administration. Toxicities that are in the opinion of the investigator(s) attributable exclusively to gemcitabine or cisplatin will not be considered DLT.
  * 7 consecutive missed doses (out of 21 doses) of enzalutamide in 21 days due to study drug related toxicity.
  * Missed day 8 dose of gemcitabine in cycle 1 will not be considered DLT.
  * Delay of greater than 3 weeks from scheduled date in initiating cycle 2 due to study drug related toxicity.
  * Discontinuation of a patient due to study drug related toxicity before completing cycle 1.
Time Frame: Up to 6 months
Population: All participants in Dose Escalation arm.
Measure: Number; unit: mg
Arm/Group | Dose Escalation
Number analyzed (Participants) | 6
mg | 160

2. Secondary Outcome: Overall Response Rate (ORR): Complete Response (CR) + Partial Response (PR)
Description: Dose Expansion. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 6 months
Population: All participants evaluable at time of analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation: Level 2 Dose: Dose Escalation - Level 2 dose of 160 mg enzalutamide (orally) with standard dose of cisplatin and gemcitabine via intravenous (IV).
- Dose Expansion: Dose Expansion: Enzalutamide at MTD (160 mg) with standard doses of cisplatin and gemcitabine.
Arm/Group | Dose Escalation: Level 1 Dose | Dose Escalation: Level 2 Dose | Dose Expansion
Number analyzed (Participants) | 3 | 3 | 4
Participants
  Partial Response | 0 | 3 | 1
  Progressive Disease | 1 | 0 | 0
  Stable Disease | 1 | 0 | 1
  Complete Response | 0 | 0 | 1
  Not Evaluable | 1 | 0 | 1

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Dose Expansion. PFS is defined as the time from randomization until objective tumor progression or death. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: 14 months
Population: All Participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation: Level 1 Dose | Dose Escalation: Level 2 Dose | Dose Expansion
Number analyzed (Participants) | 3 | 3 | 4
months | 3.81 [1.45 to 4.14] | 14.63 [13.71 to 15.88] | 7.68 [6.25 to 10.03]

4. Secondary Outcome: Overall Survival (OS)
Description: Dose Expansion. Overall survival is defined as the time from randomization until death from any cause, and is measured in the intent-to-treat population.
Time Frame: Up to 24 Months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Dose Escalation: Level 2 Dose: Dose Escalation: Level 2 dose of 160 mg enzalutamide (orally) with standard dose of cisplatin and gemcitabine via intravenous (IV).
Arm/Group | Dose Escalation: Level 1 Dose | Dose Escalation: Level 2 Dose | Dose Expansion
Number analyzed (Participants) | 3 | 3 | 4
months | 4.14 [3.81 to 10.59] | 14.63 [13.71 to 22.09] | 10.03 [6.25 to 20.05]

ADVERSE EVENTS:
Time Frame: 2 years, 7 months
Description: Patient deaths listed in "all cause mortality" occurred after the Adverse Event reporting period, but within the Overall Survival follow-up period.
Groups:
- Dose Escalation: Dose Level 1: Dose Escalation: Level 1 dose of 80 mg enzalutamide (orally), with standard doses of cisplatin and gemcitabine via intravenous (IV).
Arm/Group | Dose Escalation: Dose Level 1 | Dose Escalation: Level 2 Dose | Dose Expansion
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 2/4
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 3/4
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: Dose Level 1 (N=3) | Dose Escalation: Level 2 Dose (N=3) | Dose Expansion (N=4)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: Dose Level 1 (N=3) | Dose Escalation: Level 2 Dose (N=3) | Dose Expansion (N=4)
Fatigue (General disorders) | 3 (4) | 3 (5) | 3 (8)
Edema limbs (General disorders) | 1 (2) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 3 (3) | 3 (23) | 3 (13)
Lymphocyte count decreased (Investigations) | 0 (0) | 3 (12) | 2 (5)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (12) | 2 (5)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (5) | 2 (4)
Creatinine increased (Investigations) | 1 (3) | 2 (9) | 1 (2)
Weight loss (Investigations) | 2 (3) | 1 (3) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 3 (6) | 1 (7)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (3) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 2 (7) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 3 (7) | 2 (4) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (5) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 2 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (8) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (13)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (6) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 3 (19) | 4 (9)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (6) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 2 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (3) | 2 (7)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 2 (2) | 2 (4)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (2)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (3)
Hypertension (Vascular disorders) | 0 (0) | 2 (4) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Thromboembolic event (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study did not meet the anticipated accrual goal of 24 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT02300610/Prot_SAP_000.pdf